CLINICAL TRIAL: NCT01270854
Title: Normal Saline Versus Plasmalyte in Initial Resuscitation of Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200917793
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Wounds and Injuries; Multiple Trauma; Disorder of Fluid Balance
Keywords: Normal saline; Plasmalyte; Intravenous fluid; Traumatic injury; Fluid resuscitation
MeSH Terms: conditions — Wounds and Injuries; Multiple Trauma | interventions — Plasmalyte A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plasmalyte (Experimental): Administration of Plasmalyte A as the standard intravenous fluid during the first 24 hours after arrival to the hospital
  Interventions: Other: Plasmalyte A
- Normal Saline (Active Comparator): Administration of Normal Saline as the standard intravenous fluid during the first 24 hours after arrival to the hospital
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Plasmalyte A — Intravenous fluid
  Arms: Plasmalyte
Other: Normal Saline — Intravenous fluid
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to determine whether an intravenous salt solution called "Plasmalyte" causes less abnormality of the body's acid levels than a solution called "Normal Saline."

DETAILED DESCRIPTION:
Electrolyte-containing intravenous fluids are routinely administered to patients in the first few hours after acute traumatic injury. Although Normal Saline (0.9% sodium chloride) is commonly used in this setting, it causes a hyperchloremic acidosis that may exacerbate metabolic derangements that occur after acute injury. Plasmalyte A is a solution that more closely matches physiologic electrolyte levels. In this study, we will evaluate whether Plasmalyte A results in less disturbance of the base deficit 24 hours following traumatic injury than does Normal Saline.

ELIGIBILITY:
Inclusion Criteria:

* Triaged upon arrival to the hospital as severely injured
* At least 18 years of age
* Meets at least one of the following criteria:

  1. Intubated or likely to become intubated within 60 minutes of arrival at the hospital
  2. Likely to need an operation within 60 minutes of arrival
  3. Received or likely to receive a blood transfusion within 60 minutes of arrival

Exclusion Criteria:

* Greater than 60 minutes since arrival at the hospital
* Death likely within 48 hours
* Transfer from another hospital
* Pre-existing renal failure requiring dialysis
* Pregnancy
* Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in the base deficit | 24 hours after randomization
  Base deficit at 24 hours after randomization minus the base deficit at randomization

SECONDARY OUTCOMES:
Mortality | Hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Garth H. Utter, MD, Study Director — University of California, Davis; Lynette A. Scherer, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States

REFERENCES:
- [Derived] Young JB, Utter GH, Schermer CR, Galante JM, Phan HH, Yang Y, Anderson BA, Scherer LA. Saline versus Plasma-Lyte A in initial resuscitation of trauma patients: a randomized trial. Ann Surg. 2014 Feb;259(2):255-62. doi: 10.1097/SLA.0b013e318295feba. PMID 23732264